CLINICAL TRIAL: NCT03236870
Title: Postmarketing Observational Study to Evaluate the Effectiveness and Patient-Reported Outcome of Adalimumab in Patients With Moderate to Severe Plaque Psoriasis in China
Brief Title: A Study to Evaluate the Effectiveness and Patient-Reported Outcome of Adalimumab in Patients With Moderate to Severe Plaque Psoriasis in China
Acronym: ADAPT
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-986
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Psoriasis
Keywords: psoriasis; effectiveness; safety; adalimumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with moderate to severe plaque psoriasis in China: Participants with moderate to severe plaque psoriasis in China receiving adalimumab in daily clinical practice.

SUMMARY:
The objective of this non-interventional, observational study is to assess the effectiveness and patient reported outcome of adalimumab in patients with moderate to severe psoriasis in real world clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:

* Participant who is in compliance with eligibility for adalimumab based on the local label;
* Moderate to severe plaque psoriasis patients eligible to use adalimumab according to the local label without any contraindication
* Patients have signed the authorization (or informed consent where applicable) to disclose and use personal health information after been prescribed with adalimumab.

Exclusion Criteria:

* Patients who are pregnant or breast feeding at enrolment or wish to become pregnant during the following adalimumab treatment and within 150 days since adalimumab discontinuation;
* Patients in any psoriasis related clinical trial at the time of enrolment, at baseline or at any point during the study follow-up;
* Patients with active tuberculosis or other severe infections (e.g. sepsis and opportunistic infections) as well as moderate to severe cardiac insufficiency.
* Patients with difficulties for adequately reading, understanding and completing patient questionnaires.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate to severe plaque psoriasis in China
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving at least a 75% reduction in Psoriasis Area Severity Index (PASI) relative to the baseline PASI score | At Week 12
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination.

SECONDARY OUTCOMES:
Change from Baseline in Dermatology Life Quality Index (DLQI) | From Week 0 to Week 12
  The DLQI is a self administered short, simple and practical dermatology-specific quality of life (QoL) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (15):
- China (15):
  - The First Affiliated Hospital /ID# 171398, Hefei, Anhui
  - Guangzhou 1st Muni People Hosp /ID# 208858, Guangzhou, Guangdong
  - Ruijin Hospital, Shanghai Jiaotong /ID# 169833, Shanghai, Shanghai Municipality
  - Traditional Chinese Medical Hospital of xinjiang uygur autonomous region /ID# 209183, Ürümqi, Xinjiang
  - The Second Affiliated Hospital /ID# 169842, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital /ID# 169834, Jianggan Hangzhou, Zhejiang
  - Peking University 3rd Hospital /ID# 213443, Beijing
  - Dermatology Hospital of southe /ID# 169830, Guangzhou
  - 2nd Aff. Hosp Harbin Med Univ /ID# 169827, Haerbin
  - Shandong Provincial Hospital /ID# 169841, Jinan
  - The Tenth People's Hospital of /ID# 169831, Shanghai
  - The First Affiliated Hospital of Shantou University Medical College /ID# 209260, Shantou
  - The 7th People's Hospital of Shenyang /ID# 169829, Shenyang
  - Shenzhen Hospital of Southern /ID# 169828, Shenzhen
  - Jing Tai Tianjin Hospital Co.,Ltd /ID# 208201, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/adalimumab_P15-986.pdf